CLINICAL TRIAL: NCT01988298
Title: Ibuprofen Versus Acetaminophen in Women With Severe Pre-eclampsia After Vaginal Delivery.
Brief Title: Nonsteroidal Antiinflammatory Drugs in Women With Postpartum Pre-eclampsia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other)
Responsible Party: Principal Investigator, Paulino Vigil-De Gracia, Gynecology and obstetric, investigator and teaching proffesor, Complejo Hospitalario Dr. Arnulfo Arias Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Complejoh 02
Record Dates: First submitted 2013-10-31; First posted 2013-11-20 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental): Experimental: Ibuprofen 400 mg each 8 hours for 2-3 days.
  Interventions: Drug: Ibuprofen
- Acetaminophen (Active Comparator): Acetaminophen 1 g oral each 6 hours, 2-3 days.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 400 mg each 8 hours
  Other Names: Ibuprofen in pre-eclampsia
  Arms: Ibuprofen
Drug: Acetaminophen — Control group
  Other Names: Acetaminophen in pre-eclampsia
  Arms: Acetaminophen

SUMMARY:
Hypertensive disorders of pregnancy are a major cause of maternal mortality and morbidity, especially in developing countries. Postpartum hypertension can be related to persistence of gestational hypertension, preeclampsia, or preexisting chronic hypertension, or it could develop de novo secondary to other causes. The available data in the medical literature have primarily focused on antenatal and peripartum management. There are few data regarding the evaluation in women who are diagnosis with postpartum hypertension. Some medications that cause vasoconstriction are often used for pain relief, in women having perineal lacerations, episiotomy, or cesarean delivery. Such women usually require large doses of nonsteroidal antiinflammatory drugs that are associated with vasoconstriction and sodium and water retention, this drugs can result in severe hypertension.

The purpose of this study is to evaluate maternal postpartum hypertension in women with severe preeclampsia treated with nonsteroidal antiinflammatory drugs or acetaminophen.

DETAILED DESCRIPTION:
Our objective is evaluate Ibuprofen or acetaminophen used for pain during the postpartum period in women with severe pre-eclampsia. We include only women with vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

Vaginal delivery severe pre-eclampsia severe gestational hypertension aggregate pre-eclampsia

Exclusion Criteria:

sensitivities to ibuprofen cesarean delivery

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
level of postpartum hypertension | levels of hypertension up to 4 days post paertum
  hypertension during the postpartum using acetaminophen or nonsteroidal antiinflammatory

SECONDARY OUTCOMES:
complications | complications during the postpartum period (4 days)
  Renal failure, symptoms, bleeding

OTHER OUTCOMES:
convulsions | maternal complicactions for 4 days postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Paulino Vigil-De Gracia, MD, Study Chair — Complejo Hospitalario Caja de Seguro social
Locations (1):
- Paulino Vigil-De Gracia, Panama City, Provincia de Panamá, Panama